CLINICAL TRIAL: NCT04013672
Title: Phase II Study of Pembrolizumab Plus SurVaxM for Glioblastoma at First Recurrence
Brief Title: Study of Pembrolizumab Plus SurVaxM for Glioblastoma at First Recurrence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David Peereboom (Other)
Responsible Party: Sponsor-Investigator, David Peereboom, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE6318
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — pembrolizumab; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; montanide ISA 51

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A - Have not received immunotherapy (Experimental): Arm A is patients with first recurrence of glioblastoma who have failed prior chemotherapy and radiation but have not received any immunotherapy.
  Interventions: Drug: Pembrolizumab; Drug: SurVaxM; Drug: Sargramostim; Drug: Montanide ISA 51
- Arm B - Have failed prior anti-PD1 therapy (Experimental): Arm B is an exploratory arm of 10 patients who have failed prior anti-PD1 therapy.
  Interventions: Drug: Pembrolizumab; Drug: SurVaxM; Drug: Sargramostim; Drug: Montanide ISA 51

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg IV every 3 weeks
Drug: SurVaxM — 500 mcg per dose, dosed every two weeks for 4 doses and then every 3 months
  Other Names: SVN53-67; M57-KLH
Drug: Sargramostim — 100 mcg per dose, dosed every two weeks for 4 doses and then every 3 months
  Other Names: GM-CSF
Drug: Montanide ISA 51 — 1 ml per dose dosed every two weeks for 4 doses and then every 3 months

SUMMARY:
The main purpose of this study is to assess the clinical activity of Pembrolizumab and SurVaxM in participants with recurrent glioblastoma.

DETAILED DESCRIPTION:
Primary objective: Assess clinical activity of Pembrolizumab and SurVaxM in participants with recurrent glioblastoma using progression free survival at 6 months (PFS-6).

Secondary objective: : Assess safety and tolerability of Pembrolizumab and SurVaxM in participants with recurrent glioblastoma.

This is a Phase II study of two arms in participants with recurrent glioblastoma. Arm A will include participants with first recurrence of glioblastoma who have failed prior chemotherapy and radiation but have not received any immunotherapy. Arm B is an exploratory arm of 10 participants who have failed prior anti-PD1 therapy.

All patients will receive the study drug combination consisting of SurVaxM and pembrolizumab (PEM) with no randomization, stratification or dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of World Health Organization Grade IV glioma (glioblastoma or gliosarcoma)
* Previous first line treatment with at least radiotherapy with or without temozolomide
* Documented first recurrence of GBM by diagnostic biopsy or contrast enhanced magnetic resonance imaging (MRI) performed within 21 days of randomization per RANO criteria.
* If first recurrence of GBM is documented by MRI, an interval of at least 12 weeks after the end of prior radiation therapy is required unless there is either:

  -- Histopathologic confirmation of recurrent tumor, or

  -- New enhancement on MRI outside of the radiotherapy treatment field
* Karnofsky performance status of 70 or higher or ECOG 0-2
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study drug.
* Previous treatment with anti PD1 will be allowed only in the exploratory arm
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archive tissue
* Screening/Baseline laboratory values must meet the following criteria (laboratory value):

  --Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

  ---Hematological system:
  * Absolute neutrophil count (ANC) ≥1500/uL
  * Platelets ≥100 000/µL
  * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L (Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.)

    ---Renal system:
  * Creatinine OR Measured or calculated (Creatinine clearance (CrCl) should be calculated per institutional standard) creatinine clearance (GFR can also be used in place of creatinine or CrCl): ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN

    ---Hepatic system:
  * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
  * AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)

    --- Coagulation system:
  * International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT): ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* Male participants:

  --A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period.
* Female participants:

  * A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

    * Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
    * A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 180 days after the last dose of study treatment.

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has received prior therapy with an anti-PD-1 (except in the exploratory arm), anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to (randomization /allocation).

  * Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.
  * Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

  --Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 2 mg daily of dexamethasone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Patients that likely to have the potential risk of cerebral edema due to inflammation related to SurVaxM and pembrolizumab and will exclude patients with > 1 cm midline shift on imaging. Patients ust not have cerebral edema requiring more than 2 mg of daily of dexamethasone equivalent.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* More than one recurrence of GBM
* Presence of extracranial metastatic or leptomeningeal disease
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy .Has a known history of Human Immunodeficiency Virus (HIV). No HIV testing is required
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Peereboom, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share main findings of the clinical study report (CSR)
Supporting Information: CSR

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A - Have Not Received Immunotherapy | Arm B - Have Failed Prior Anti-PD1 Therapy
Started | 41 | 0
Completed | 32 | 0
Not Completed | 9 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Death | 1 | 0
Not completed — Physician Decision | 5 | 0

BASELINE CHARACTERISTICS:
Population: Exploratory arm was not conducted
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Have Not Received Immunotherapy | Arm B - Have Failed Prior Anti-PD1 Therapy | Total
Number analyzed (Participants) | 41 | 0 | 41
Age, Customized [Count of Participants; unit: Participants]
  20-29 | 1 |  | 1
  30-39 | 3 |  | 3
  40-49 | 5 |  | 5
  50-59 | 15 |  | 15
  60-69 | 11 |  | 11
  70-79 | 6 |  | 6
  80-89 | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 |  | 18
  Male | 23 |  | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 1
  Not Hispanic or Latino | 37 |  | 37
  Unknown or Not Reported | 3 |  | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 38 |  | 38
  More than one race | 0 |  | 0
  Unknown or Not Reported | 3 |  | 3
MGMT_Methylation [Count of Participants; unit: Participants] — MGMT methylation = tumor methylation status of methyl guanine methyl transferase, a prognostic factor in GBM Population: Only 40 analyzed for this measure for MGMT_Methylation
  Participants
    number analyzed (Participants) | 40 | 0 | 40
    No | 24 |  | 24
    Unknown | 1 |  | 1
    Yes | 15 |  | 15
Number_of_Prior_Surgeries [Count of Participants; unit: Participants]
  1 | 31 |  | 31
  2 | 9 |  | 9
  3 | 1 |  | 1
Temodar_with_Radiation__Concurre [Count of Participants; unit: Participants]
  No | 5 |  | 5
  Yes | 36 |  | 36
kps_bs [Count of Participants; unit: Participants] — KPS_BS = Karnofsky performance score at baseline
  The Karnofsky Performance Status (KPS) assesses a patient's ability to perform daily activities, predicting prognosis and suitability for clinical trials. Scores range from 0 to 100.
  100: Normal 90: Minor symptoms 80: Some effort needed 70: Can self-care, but not normal activities 60: Needs occasional help 50: Needs considerable help 40: Requires special care 30: Severely ill; needs hospitalization 20: Very ill; active support needed 10: Moribund; rapidly worsening 0: Dead
  Participants
    70 | 9 |  | 9
    80 | 19 |  | 19
    90 | 13 |  | 13
Temodar_Alone__Adjuvant__ [Count of Participants; unit: Participants]
  No | 8 |  | 8
  Yes | 33 |  | 33
Clinical_Trial_given_drugs [Count of Participants; unit: Participants]
  No/Unknown | 19 |  | 19
  Yes | 22 |  | 22

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Assess clinical activity of Pembrolizumab and SurVaxM in patients with recurrent glioblastoma using PFS at 6 months (PFS-6)
Time Frame: 6 months from start of treatment
Population: Exploratory arm was not conducted
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A - Have Not Received Immunotherapy | Arm B - Have Failed Prior Anti-PD1 Therapy
Number analyzed (Participants) | 41 | 0
percentage of participants | 34.5 [19.8 to 49.6] |

2. Secondary Outcome: Safety and Tolerability of Pembrolizumab and SurVaxM as Measure by CTCAE v 5 Grading as Per NCI
Description: Safety and tolerability of Pembrolizumab and SurVaxM in patients with recurrent glioblastoma measured on ongoing basis with CTCAE v 5 grading as per NCI. Grade 1-2 and 3-5 events will be recorded and reported.
Time Frame: up to 1 year from enrollment
Population: Exploratory arm was not conducted
Measure: Number; unit: Events
Arm/Group | Arm A - Have Not Received Immunotherapy | Arm B - Have Failed Prior Anti-PD1 Therapy
Number analyzed (Participants) | 41 | 0
Events
  Number of CTCAE V5 Events with Grades 1-2 | 481 |
  Number of CTCAE V5 Events with Grades 3-5 | 107 |
  Possible AEs related to Pembrolizumab | 43 |
  Probable AEs related to Pembrolizumab | 6 |
  Unlikely AEs related to Pembrolizumab | 31 |
  Unrelated AEs to Pembrolizumab | 508 |
  Definite AEs related to SurVaxM | 6 |
  Possible AEs related to SurVaxM | 25 |
  Probable AEs related to SurVaxM | 38 |
  Unlikely AEs related to SurVaxM | 67 |
  Unrelated AEs to SurVaxM | 452 |
  Definite AEs related to disease | 39 |
  Possible AEs related to disease | 90 |
  Probable AEs related to disease | 104 |
  Unlikely AEs related to disease | 43 |
  Unrelated AEs to disease | 312 |

ADVERSE EVENTS:
Time Frame: Day 1 of treatment until 30 days after patient went off study, upto 19.7 months
Description: Exploratory arm was not conducted
Arm/Group | Arm A - Have Not Received Immunotherapy | Arm B - Have Failed Prior Anti-PD1 Therapy
All-Cause Mortality (participants affected / at risk) | 1/41 | 0/0
Serious Adverse Events (participants affected / at risk) | 22/41 | 0/0
Other Adverse Events (participants affected / at risk) | 41/41 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - Have Not Received Immunotherapy (N=41) | Arm B - Have Failed Prior Anti-PD1 Therapy (N=0)
Cardiac arrest (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Disease progression (General disorders) | 3 | 0
Edema limbs (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Fever (General disorders) | 1 | 0
Gait disturbance (General disorders) | 2 | 0
Injection site reaction (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 3 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Cognitive disturbance (Nervous system disorders) | 5 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Dysphasia (Nervous system disorders) | 2 | 0
Edema cerebral (Nervous system disorders) | 6 | 0
Facial muscle weakness (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 3 | 0
Lethargy (Nervous system disorders) | 1 | 0
Muscle weakness left-sided (Nervous system disorders) | 4 | 0
Muscle weakness right-sided (Nervous system disorders) | 2 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 3 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 6 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Agitation (Nervous system disorders) | 1 | 0
Anxiety (Nervous system disorders) | 1 | 0
Confusion (Nervous system disorders) | 1 | 0
Personality change (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Thromboembolic event (Vascular disorders) | 3 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Have Not Received Immunotherapy (N=41) | Arm B - Have Failed Prior Anti-PD1 Therapy (N=0)
alt increased (Investigations) | 8 | 0 (0)
anc decreased (Investigations) | 3 | 0 (0)
anc increased (Investigations) | 6 | 0 (0)
anemia (Investigations) | 2 | 0 (0)
leukocytosis (Investigations) | 1 | 0 (0)
platelet decreased (Investigations) | 6 | 0 (0)
wbc decreased (Investigations) | 4 | 0 (0)
wbc increased (Investigations) | 6 | 0 (0)
angina (Cardiac disorders) | 1 | 0 (0)
cardiac arrest (Cardiac disorders) | 1 | 0 (0)
facial flushing (Cardiac disorders) | 1 | 0 (0)
hypertension (Cardiac disorders) | 3 | 0 (0)
hypotension (Cardiac disorders) | 3 | 0 (0)
palpitations (Cardiac disorders) | 1 | 0 (0)
pulmonary embolism (Cardiac disorders) | 2 | 0 (0)
tachycardia (Cardiac disorders) | 1 | 0 (0)
thrombocytosis (Cardiac disorders) | 6 | 0 (0)
ear pain (Ear and labyrinth disorders) | 2 | 0 (0)
hearing loss (Ear and labyrinth disorders) | 1 | 0 (0)
vertigo (Ear and labyrinth disorders) | 1 | 0 (0)
decreased t3 (Investigations) | 2 | 0 (0)
decreased t4 (Investigations) | 1 | 0 (0)
decreased tsh (Investigations) | 2 | 0 (0)
hyperthyroidism (Investigations) | 2 | 0 (0)
hypophysitis (Investigations) | 1 | 0 (0)
hypothyroidism (Investigations) | 4 | 0 (0)
increased t4 (Investigations) | 1 | 0 (0)
increased tsh (Investigations) | 2 | 0 (0)
blurry vision (Eye disorders) | 2 | 0 (0)
cataracts (Eye disorders) | 1 | 0 (0)
decreased depth perception (Eye disorders) | 1 | 0 (0)
diplopia (Eye disorders) | 1 | 0 (0)
eye irritation (Eye disorders) | 1 | 0 (0)
peripheral vision (Eye disorders) | 1 | 0 (0)
photophobia (Eye disorders) | 1 | 0 (0)
blisters lip (General disorders) | 1 | 0 (0)
chills (General disorders) | 3 | 0 (0)
cough (General disorders) | 2 | 0 (0)
decreased appetite (General disorders) | 4 | 0 (0)
dry mouth (General disorders) | 2 | 0 (0)
extravastion (General disorders) | 1 | 0 (0)
extremity pain (General disorders) | 2 | 0 (0)
face edema (General disorders) | 1 | 0 (0)
falls (General disorders) | 18 | 0 (0)
fatigue (General disorders) | 17 | 0 (0)
fever (General disorders) | 2 | 0 (0)
flu symptoms (General disorders) | 2 | 0 (0)
generalized edema (General disorders) | 1 | 0 (0)
heat intolerance (General disorders) | 1 | 0 (0)
infection (General disorders) | 3 | 0 (0)
insomnia (General disorders) | 6 | 0 (0)
lethargy (General disorders) | 2 | 0 (0)
limbs edema (General disorders) | 3 | 0 (0)
oral (General disorders) | 2 | 0 (0)
other (General disorders) | 1 | 0 (0)
pain (General disorders) | 1 | 0 (0)
rib pain (General disorders) | 1 | 0 (0)
weight loss (General disorders) | 1 | 0 (0)
abdominal bloating (Gastrointestinal disorders) | 1 | 0 (0)
canker sore (mouth pain) (Gastrointestinal disorders) | 1 | 0 (0)
checkpoint inhibitor hepatitis (Gastrointestinal disorders) | 1 | 0 (0)
constipation (Gastrointestinal disorders) | 4 | 0 (0)
diarrhea (Gastrointestinal disorders) | 8 | 0 (0)
dysphagia (Gastrointestinal disorders) | 6 | 0 (0)
gas (belching) (Gastrointestinal disorders) | 1 | 0 (0)
gerd (Gastrointestinal disorders) | 1 | 0 (0)
investigations (Gastrointestinal disorders) | 1 | 0 (0)
nausea (Gastrointestinal disorders) | 8 | 0 (0)
vomiting (Gastrointestinal disorders) | 4 | 0 (0)
infection of unknown etiology (Infections and infestations) | 1 | 0 (0)
lung infection (Infections and infestations) | 2 | 0 (0)
possible sepsis (Infections and infestations) | 1 | 0 (0)
abnormal electrocytes (Investigations) | 8 | 0 (0)
adrenal insufficiency (Investigations) | 1 | 0 (0)
alkaline phosphatase increased (Investigations) | 1 | 0 (0)
allergic reaction (Investigations) | 1 | 0 (0)
ast increased (Investigations) | 9 | 0 (0)
bruising (generalized) (Investigations) | 1 | 0 (0)
death (Investigations) | 8 | 0 (0)
hyperglycemia (Investigations) | 6 | 0 (0)
multisystem organ failure (Investigations) | 1 | 0 (0)
other (Investigations) | 1 | 0 (0)
decreased appetite (Metabolism and nutrition disorders) | 2 | 0 (0)
decreased phosphorus (Metabolism and nutrition disorders) | 1 | 0 (0)
hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 (0)
ankle swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 (0)
decreased mobility (Musculoskeletal and connective tissue disorders) | 1 | 0 (0)
extremity pain (Musculoskeletal and connective tissue disorders) | 1 | 0 (0)
musculoskeletal (Musculoskeletal and connective tissue disorders) | 22 | 0 (0)
neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 (0)
paresthesia (Musculoskeletal and connective tissue disorders) | 14 | 0 (0)
neoplasms benign or malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 (0)
altered sense of smell (Nervous system disorders) | 1 | 0 (0)
aphasia (Nervous system disorders) | 4 | 0 (0)
cerebral edema (Nervous system disorders) | 7 | 0 (0)
cognitive disturbance (Nervous system disorders) | 19 | 0 (0)
decreased consciousness (Nervous system disorders) | 2 | 0 (0)
dizziness (Nervous system disorders) | 4 | 0 (0)
edema cerebral (Nervous system disorders) | 2 | 0 (0)
fine motor skills change (Nervous system disorders) | 2 | 0 (0)
headache (Nervous system disorders) | 18 | 0 (0)
intermittent metallic taste (Nervous system disorders) | 1 | 0 (0)
memory loss (Nervous system disorders) | 4 | 0 (0)
mental or emotional change (Nervous system disorders) | 14 | 0 (0)
numbness (Nervous system disorders) | 3 | 0 (0)
paresthesia (Nervous system disorders) | 14 | 0 (0)
seizure (Nervous system disorders) | 11 | 0 (0)
sensation changes (Nervous system disorders) | 2 | 0 (0)
spasticity (Nervous system disorders) | 1 | 0 (0)
speech changes (Nervous system disorders) | 2 | 0 (0)
tremor (Nervous system disorders) | 4 | 0 (0)
cpk increased (Renal and urinary disorders) | 1 | 0 (0)
creatinine increased (Renal and urinary disorders) | 4 | 0 (0)
glucosuria (Renal and urinary disorders) | 3 | 0 (0)
hemaglobinuria (Renal and urinary disorders) | 1 | 0 (0)
proteinuria (Renal and urinary disorders) | 18 | 0 (0)
urinary frequency change (Renal and urinary disorders) | 4 | 0 (0)
urinary s/s (Renal and urinary disorders) | 1 | 0 (0)
urinary tract infection (Renal and urinary disorders) | 1 | 0 (0)
urinary urgency (Renal and urinary disorders) | 3 | 0 (0)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
epistaxis (nose bleed) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
pleural effusion (left) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
rhinnorhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
throat mucous (postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 (0)
generalized rash (Skin and subcutaneous tissue disorders) | 1 | 0 (0)
injection site reaction (Skin and subcutaneous tissue disorders) | 19 | 0 (0)
night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 (0)
photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0 (0)
pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 4 | 0 (0)
swelling at craniotomy site (Skin and subcutaneous tissue disorders) | 1 | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT04013672/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT04013672/ICF_001.pdf